CLINICAL TRIAL: NCT00746473
Title: Assessment of Cytokine Values in Serum and by Specific cDNA Amplification and Detection Using RT-PCR in HIV-1 Infected Individuals With and Without Highly Active Anti-Retroviral Therapy (HAART)
Brief Title: Assessment of Cytokine Values in Serum and by RT-PCR in HIV-1 Individuals With and Without HAART
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Sergio Muller, Faculdade de Medicina de Botucatu - Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-12
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: 15 HIV-1 infected individuals, with or without AIDS, who had never received ARV. These patients had not yet been indicated for ARV, or had had HIV-1 infection diagnosed a few days before inclusion in this study.
- 2: 27 HIV-1 infected individuals, sick or not, on ARV treatment, five with two nucleoside/nucleotide reverse transcriptase inhibitors (NRTI) and one nonnucleoside reverse transcriptase inhibitor (NNRTI), and 22 on HAART with two NRTI, or one NRTI and one NNRTI, and one protease inhibitor (PI), and VL equal to or greater than 50 copies of plasma RNA/mL.
  Treatment duration in this group varied between three and 145 months (mean 53.62 months; median 42 months).
- 3: 31 HIV-1 infected individuals on ARV treatment, 16 on HAART with two NRTI, or one NRTI and one NNRTI, and one PI, and 15 with two NRTI and one NNRTI. All G3 patients had undetectable VL for at least the past 6 months. Treatment in this group varied between five to 108 months (mean 48.13 months; median 42 months).
- 4: 20 blood donors without clinical complaints and negative for anti-HIV-1/2 antibodies. None of them showed any sign of disease.

SUMMARY:
A cross-sectional study was performed on HIV-1 infected individuals with or without antiretroviral treatment. 73 HIV-1 infected individuals were divided into three groups: G1= 15 infected individuals with or without AIDS who never received ARV; G2= 27 patients on HAART, and plasma HIV-1 RNA viral load (VL) equal or greater than 50 copies/mL and G3= 31 patients on HAART with undetectable VL for at least the past 6 months and a fourth group G4= 20 individuals chosen between blood donors without any disease sign and with negative HIV serum tests (control group). Serum cytokine levels pg/mL (ELISA) and specific mRNA expression by RT-PCR were performed on all four groups for TNF-a, IL-2, INF-g, IL-4 and IL-10. All patients were submitted to VL determination and CD4+ and CD8+T lymphocyte counts. Results analysis showed a significant comparison between groups for both methods and association between them (>80% - r2>0.80) with only one exception, in the individuals of control group, for IL-2 by ELISA determination. The cytokine profile for both methods and three patient groups was mature Th-0. The behavior of IL-2 and INF-g must be emphasized with the consequent expression on dominant Th profile. Both methods showed low IL-2 and elevated mean INF-g values in the three patient groups.

DETAILED DESCRIPTION:
A cross-sectional study was performed on HIV-1 infected individuals with or without antiretroviral treatment (ARV) at the AIDS Day-Hospital, Botucatu School of Medicine, Unesp. Between August 2004 and October 2005, 73 HIV-1 infected individuals were divided into three groups: G1= 15 infected individuals with or without AIDS who never received ARV; G2= 27 patients on HAART, and plasma HIV-1 RNA viral load (VL) equal or greater than 50 copies/mL and G3= 31 patients on HAART with undetectable VL for at least the past 6 months and a fourth group G4= 20 individuals chosen between blood donors without any disease sign and with negative HIV serum tests (control group). Serum cytokine levels pg/mL (ELISA) and specific mRNA expression by RT-PCR were performed on all four groups for TNF-a, IL-2, INF-g, IL-4 and IL-10. All patients were submitted to VL determination and CD4+ and CD8+T lymphocyte counts. Results analysis showed a significant comparison between groups for both methods and association between them (>80% - r2>0.80) with only one exception, in the individuals of control group, for IL-2 by ELISA determination. The cytokine profile for both methods and three patient groups was mature Th-0. The behavior of IL-2 and INF-g must be emphasized with the consequent expression on dominant Th profile. Both methods showed low IL-2 and elevated mean INF-g values in the three patient groups. Several authors have recently drawn attention to the substantial apoptosis of infected and non infected CD4+T cells, mainly during primary infection, persisting only in those with INF-g phenotype producer and not IL-2.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection

Exclusion Criteria:

* no HIV infection

Ages: 22 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All 73 HIV-1 infected individuals were submitted to full clinical observation including associated opportunistic diseases at time of blood collection for cytokine detection.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2004-08; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domingos A Meira, PhD, MD, Principal Investigator — Faculdade de Medicina de Botucatu, Unesp
Locations (1):
- SAE e Hospital Dia de Aids, Botucatu, São Paulo, Brazil